CLINICAL TRIAL: NCT01644825
Title: MITO-11: A Randomized Multicentre Phase II Trial With Pazopanib and Weekly Paclitaxel vs Weekly Paclitaxel in Platinum Resistant or Refractory Ovarian Cancer
Brief Title: Weekly Paclitaxel With or Without Pazopanib in Platinum Resistant or Refractory Ovarian Cancer
Acronym: MITO-11
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MITO-11; 2009-016151-21 (EudraCT Number)
Record Dates: First submitted 2012-07-17; First posted 2012-07-19 (Estimated); Last update posted 2018-04-09 (Actual); Status verified 2018-04

CONDITIONS: Ovarian Cancer
Keywords: platinum resistant; platinum refractory
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Paclitaxel; pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- paclitaxel and pazopanib (Experimental)
  Interventions: Drug: paclitaxel; Drug: pazopanib
- paclitaxel (Active Comparator)
  Interventions: Drug: paclitaxel

INTERVENTIONS:
Drug: paclitaxel — 80 mg/m2 IV days 1, 8, 15 every 28 days
Drug: pazopanib — orally, 800 mg orally daily
  Arms: paclitaxel and pazopanib

SUMMARY:
The purpose of this study is to evaluate the safety and activity of adding pazopanib to weekly chemotherapy with paclitaxel for patients with ovarian cancer that is resistant or refractory to treatment with platinum based therapy.

ELIGIBILITY:
Inclusion Criteria:

* Cytologic / histologic diagnosis of stage IC-IV ovarian cancer
* Disease progressed during first line chemotherapy or disease relapsed within 6 months after the last platinum treatment
* Disease evaluable by RECIST or Ca 125 GCIG criteria
* No residual peripheral neurotoxicity from previous chemotherapy treatment
* PS 0-1
* Aged at least 18 and not greater than 75 years.
* Life expectancy of at least 3 months
* Able to swallow and retain oral medication
* Written informed consent prior to performance of study specific procedures or assessments
* Ability and willingness to comply with treatment and follow up assessments and procedures

Exclusion Criteria:

· • Previous or concomitant malignant neoplasia (not including basocellular or spinocellular skin carcinoma or in-situ carcinoma of the uterine cervix, provided they are being adequately treated)

* Previous treatment with weekly paclitaxel
* More than 2 previous chemotherapy treatments
* Serious heart disease, including heart failure, atrioventricular block of any degree, serious arrhythmia or history of any one or more of the following cardiovascular conditions within the past 6 months: cardiac angioplasty or stenting, myocardial infarction, unstable angina, symptomatic peripheral vascular disease, coronary artery by-pass graft surgery, class II, III or IV congestive heart failure as defined by the New York Heart Association (NYHA)
* Hemoglobin < 9 g/dL, neutrophils < 1500/mm3, platelets < 100000/mm3
* Impairment of renal function (patients should have 2 functioning kidneys): creatinine 1.5 times the upper normal limit - UNL; calculated creatinine clearance < 50 mL/min; urine protein to creatinine ratio > or = 1: then, a 24-hour urine protein must be assessed and subject must have a 24-hour urine protein value <1gr to be eligible
* Impairment of liver function (SGOT or SGPT > or = 2.5 UNL, alkaline phosphatase > 2.5 ULN, total bilirubin > 1.5 times the UNL)
* Prothrombin time (PT) or international normalized ratio (INR) or activated partial thromboplastin time (PTT) > 1.2 times the UNL
* Pregnancy, breast feeding, or inadequate contraception
* Unable to discontinue prohibited medications (see protocol section 6.7)
* Clinically significant gastrointestinal abnormalities which might interfere with oral dosing, including but not limited to malabsorption syndrome, major resection of the stomach or small bowel that could affect drug absorption, active peptic ulcer disease, inflammatory bowel disease, ulcerative colitis, other gastrointestinal conditions with increased risk of perforation, history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 28 days prior to beginning study treatment, signs or symptoms of GI obstruction
* Any unstable or serious concurrent condition
* Prolongation of corrected QT interval (QTc) >480 ms
* History of cerebrovascular accident, pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months
* Macroscopic hematuria
* Major surgery or trauma within 30 days
* Hypertension uncontrolled with adequate therapy (systolic blood pressure (BP) of > or = 140mmHg, or diastolic BP of > or = 90mmHg)
* Any ongoing toxicity from prior anti-cancer therapy that is >Grade 1 and/or that is progressing in severity
* Present or suspected haemorrhagic syndromes
* Patients' inability to access the centre due to area of residence

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2010-12 (Actual); Primary Completion 2014-05 (Actual); Study Completion 2015-12-29 (Actual)

PRIMARY OUTCOMES:
progression free survival | 6 months from randomization

SECONDARY OUTCOMES:
number of patients with objective response | at 2 months and 4 months after randomization
worst grade toxicity per patient | at end of each 28 day cycle of therapy
overall survival | one year from randomization

CONTACTS AND LOCATIONS:
Overall Officials: Sandro Pignata, M.D., Ph.D., Principal Investigator — National Cancer Institute, Naples; Francesco Perrone, M.D., Ph.D., Principal Investigator — National Cancer Institute, Naples; Ciro Gallo, M.D., Ph.D., Principal Investigator — University of Campania Luigi Vanvitelli
Locations (20):
- Italy (20):
  - Osp. Regionale Mulli, Acquaviva delle Fonti
  - Ospedale San donato, Arezzo
  - A.O. G. Rummo, Benevento
  - Ospedale Bellaria, Bologna
  - Ospedale Senatore Antonio Perrino, Brindisi
  - A.O. Garibaldi Nesimadi Catania, Catania
  - Ospedale Civile di Faenza, Faenza
  - A.O.U. Arcispedale Sant'Anna di Ferrara, Ferrara
  - Ospedale Fabrizio Spaziani della ASL di Frosinone, Frosinone
  - Ospedale Umbero I, Lugo
  - Istituto Nazionale Tumori, Milan
  - A.O. Univeristaria Policlinico, Modena
  - Istituto Nazionale dei Tumori , Oncologia Medica - Dipartimento Uro-Ginecologico, Napoli
  - Seconda Universita di Napoli, Napoli
  - Ospedale Silvestrini, Perugia
  - Ospedale S. Maria delle Croci AUSL di Ravenna, Ravenna
  - A.O. Bainchi Melacrino Morelli Osp. Riuniti, Reggio Calabria
  - Ospedale degli Infermi, P.O. Ospedale Civile, Rimini
  - Policlinico Umberto I, Roma
  - Policlinico Universitario Gemelli Università Cattolica del Sacro Cuore, Roma

REFERENCES:
- [Background] Pignata S, Lorusso D, Scambia G, Sambataro D, Tamberi S, Cinieri S, Mosconi AM, Orditura M, Brandes AA, Arcangeli V, Panici PB, Pisano C, Cecere SC, Di Napoli M, Raspagliesi F, Maltese G, Salutari V, Ricci C, Daniele G, Piccirillo MC, Di Maio M, Gallo C, Perrone F; MITO 11 investigators. Pazopanib plus weekly paclitaxel versus weekly paclitaxel alone for platinum-resistant or platinum-refractory advanced ovarian cancer (MITO 11): a randomised, open-label, phase 2 trial. Lancet Oncol. 2015 May;16(5):561-8. doi: 10.1016/S1470-2045(15)70115-4. Epub 2015 Apr 14. PMID 25882986
- [Derived] Gaitskell K, Rogozinska E, Platt S, Chen Y, Abd El Aziz M, Tattersall A, Morrison J. Angiogenesis inhibitors for the treatment of epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Apr 18;4(4):CD007930. doi: 10.1002/14651858.CD007930.pub3. PMID 37185961